CLINICAL TRIAL: NCT03090997
Title: Effect of Resveratrol and Vitamin C on Insulin Resistance and Antioxidant Capacity in Postmenopausal Women. A Randomized Clinical Trial
Brief Title: Effect of Resveratrol and Vitamin C on Insulin Resistance Among Postmenopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes (Other Government)
Responsible Party: Principal Investigator, ENRIQUE REYES-Munoz MD, Clinical Professor, Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3210-10209-01-574-17
Record Dates: First submitted 2017-03-16; First posted 2017-03-27 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Postmenopausal; Insulin Resistance
Keywords: resveratrol, vitamin C, antioxidant therapy, antioxidant capacity
MeSH Terms: conditions — Insulin Resistance | interventions — Ascorbic Acid; Resveratrol

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care provider, investigator and outcomes assesor will be masking using placebo for resveratrol and vitamin C, the three groups will receive the same intervention with the use of placebo. The placebo will be prepared for the Pharmacology Department and packing and label for exclusive use into the protocol study. Any participant, care provider or investigator will know if package content vitamin C, resveratrol or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Placebo Comparator): vitamin C (500 mg/day/orally) + placebo
  Interventions: Dietary Supplement: vitamin C (500 mg / day) + placebo
- Group 2 (Placebo Comparator): resveratrol (500 mg/day/orally) + placebo
  Interventions: Dietary Supplement: resveratrol (500 mg / day) + placebo
- Group 3 (Active Comparator): vitamin C (500 mg/day/orally) + resveratrol (500 mg/day/orally)
  Interventions: Dietary Supplement: vitamin C (500 mg / day) and resveratrol (500 mg / day)

INTERVENTIONS:
Dietary Supplement: vitamin C (500 mg / day) + placebo — Adminstration of vitamin C (500 mg / day/orally) + placebo (same presentation like resveratrol)
  Arms: Group 1
Dietary Supplement: resveratrol (500 mg / day) + placebo — Adminstration of resveratrol (500 mg / day/orally) + placebo (same presentation like vitamin C)
  Arms: Group 2
Dietary Supplement: vitamin C (500 mg / day) and resveratrol (500 mg / day) — Adminstration of resveratrol (500 mg / day/orally) + vitamin C 500 mg/day/orally)
  Arms: Group 3

SUMMARY:
Hormonal and metabolic changes because of postmenopause increase body weight, central abdominal fat, alter lipid profile and insulin resistance, those factors increase the risk up to 60% to develop metabolic syndrome, diabetes and cardiovascular diseases. Because there is no efficient antioxidant therapy in postmenopausal women, this study proposes a therapy with resveratrol and vitamin C to increase the total antioxidant capacity; as well as to decrease insulin resistance and in consequence decreased the risk of diabetes, metabolic syndrome and cardiovascular disease

DETAILED DESCRIPTION:
Currently, there are not studies that demonstrate an efficient antioxidant therapy in postmenopausal women, to increase the total antioxidant capacity and to decrease insulin resistance and biochemical parameters of cardio-metabolic risk. Therefore, the aim of this study is to evaluate the effect of the co-administration of resveratrol and vitamin C on insulin resistance and antioxidant capacity by a double-blind randomized clinical trial. A population of 270 postmenopausal women will be studied, stratified into 3 groups:

Group 1: Three-month administration of vitamin C 500 mg daily + placebo Group 2: Three-month administration of resveratrol 500 mg daily + placebo Group 3: Three months administration of vitamin C 500 mg daily and resveratrol 500 mg daily as antioxidant therapy.

All participants will be monitored monthly for a period of 3 months: glucose, insulin, uric acid, Homeostatic Model Assessment (HOMA), total cholesterol (TC), triglycerides (TGC), High density lipoproteins-cholesterol (HDL- C), low density lipoproteins-cholesterol (LDL), blood pressure, body mass index (BMI). The antioxidant efficiency in erythrocytes by the quantification of antioxidant enzymes (superoxide dismutase, catalase, glutathione reductase and glutathione peroxidase), as well as total antioxidant capacity in plasma. In order to corroborate the oxidative damage, the product of the lipoperoxidation malondialdehyde and the carbonylation of proteins will be evaluated by spectrophotometric techniques before and three months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with early postmenopause according to STRAW classification.
* Insulin resistance determinated by HOMA ≥ 2.5.
* Not use of metformin, bezafibrates and / or statins, three months before enter to the study
* No indication of hormone replacement therapy.
* Sign the informed consent.

Exclusion Criteria:

* Women who present pathologies such as: Diabetes Mellitus, rheumatoid arthritis, lupus, neoplasms of any type, HIV, or kidney disease during the course of the study.
* Women who during the development of the protocol require hormone replacement therapy.
* Any type of surgical intervention during the following of the study.
* That the patient wishes to withdraw from the study.
* That the patient does not complete with 80% of adherence to the treatment

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance | HOMA at 3 months after starting the intervention in each group
  Insulin resistance measured by HOMA (Homeostatic Model Assessment)

SECONDARY OUTCOMES:
Superoxide dismutase activity | three months after starting the intervention
  Enzymatic activity measured by spectrophotometry
Catalase activity | three months after starting the intervention
  Enzymatic activity measured by spectrophotometry
Glutathione peroxidase activity | three months after starting the intervention
  Enzymatic activity measured by spectrophotometry
Glutathione reductase activity | three months after starting the intervention
  Enzymatic activity measured by spectrophotometry
Malondialdehyde | three months after starting the intervention
  Enzymatic activity measured by spectrophotometry
Carbonylation of proteins | three months after starting the intervention
  Marker of oxidative stress measured by spectrophotometry

CONTACTS AND LOCATIONS:
Overall Officials: Araceli Montoya-Estrada, PhD, Principal Investigator — Instituto Nacional de Perinatología Isidro Espinosa de los Reyes; Guillermo F Ortiz-Luna, MD, Study Chair — Instituto Nacional de Perinatología Isidro Espinosa de los Reyes
Locations (1):
- Instituto Nacional de Perinatología Isidro Espinosa de los Reyes, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Undecided